CLINICAL TRIAL: NCT00346983
Title: Pilot Study of the Effect of Pegaptanib Sodium to Prevent Worsening of Cystoid Macular Edema Following Cataract Surgery in Diabetics
Brief Title: Macugen to Prevent Worsening of Macular Edema Following Cataract Surgery in Diabetics
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling eligible subjects
Sponsor: Johns Hopkins University (Other)
Collaborators: Eyetech Pharmaceuticals (Industry)
Responsible Party: Oliver D. Schein, MD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00001385
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Cystoid Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — pegaptanib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pegaptanib sodium
- B (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Pegaptanib sodium — 0.3mg/0.1ml intravitreal injection, every 6 weeks, up to a total of 3 injections
  Other Names: Macugen
  Arms: A
Drug: Control — Sham injection, every 6 weeks, up to a total of 3 sham injections
  Arms: B

SUMMARY:
This research is being conducted to look at the effects of an intraocular drug (pegaptanib, also called Macugen) for the treatment of swelling in the retina (the light sensitive tissue in the back of the eye) that often occurs following cataract surgery in patients with diabetic eye disease. Swelling in the retina can lead to blurry vision, and Macugen may reduce this swelling. Eyedrops that decrease inflammation also may help to stop some of the swelling. We are testing this drug (pegaptanib) to see if it can decrease swelling in the retina and improve vision in patients with diabetes who are having cataract surgery.

DETAILED DESCRIPTION:
Macular edema occurs as a complication of cataract surgery in approximately 2% of all surgeries. In this condition, cystic, fluid-filled spaces develop in the outer plexiform layer of the retina resulting in a loss of vision. This condition is termed "Cystoid Macular Edema (CME)." In non-diabetics, the majority of such cases resolve spontaneously.

Diabetic macular edema (DME) is an important cause of visual disability among patients with diabetes. It is widely recognized that cataract surgery often triggers severe CME in patients with pre-existing DME. This exacerbation begins immediately following cataract surgery; and unlike in non-diabetics the edema is likely to be protracted and poorly responsive both to traditional treatments for CME (topical NSAIDS) and DME (laser photocoagulation). Fluorescein angiography, a photographic test that evaluates the blood circulation in the back of the eye, has demonstrated that both CME and DME are associated with increased permeability of retinal blood vessels.

The high rates and severity of post-cataract surgery CME in diabetic patients with DME render this population ideal for the study of potential agents to reduce the rate and severity of this condition (i.e., post-cataract surgery CME). Recent studies have shown that vascular endothelial growth factor (VEGF) plays a major role in vessel permeability. Pegaptanib (Macugen) is an FDA-approved drug for wet AMD. Pegaptanib is a selective VEGF antagonist that blocks the effects of VEGF; therefore pegaptanib might decrease vessel permeability and possibly decrease the incidence and severity of CME. We plan to conduct a controlled pilot study to investigate the effects of pegaptanib (up to 3 treatments of pegaptanib given prior to cataract surgery and as often as every 6 weeks for up to 12 weeks after cataract surgery) in diabetic patients with pre-existing DME who are undergoing cataract surgery and who are, therefore, at very high risk for development of CME. Should the pilot study indicate a potential benefit of pegaptanib in this setting, a larger, fully powered clinical trial will be proposed. An effective treatment or preventive measure for post-cataract surgery macular edema in patients with diabetic retinopathy would offer benefit to a large patient population nationally that is at high risk of vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 years or older) with diabetes mellitus
* Best corrected visual acuity worse than 20/40 but no worse than 20/800 in the study eye
* Best corrected visual acuity better than or equal to 20/800 in the fellow eye
* DME in the study eye (eye scheduled to undergo cataract surgery) as documented on OCT as a center point thickness of at least 250 microns no more than 3 weeks prior to cataract surgery
* No prior laser photocoagulation in the study eye for at least 4 months prior to cataract surgery
* Women of child-bearing potential who are interested in participating in this study will use two effective forms of contraception prior to initiation of pegaptanib and then throughout the remainder of the study. For women of childbearing potential, results from a urine pregnancy test will be obtained prior to each injection with pegaptanib. Urine samples will be disposed of after the test is performed.

Exclusion Criteria:

* History of intravitreal steroid (triamcinolone) injection into the study eye within 4 months prior to cataract surgery
* Macular edema due to non-diabetic etiologies such as vein occlusion
* Retinal diseases that preclude evaluation of the macula for edema (e.g., macular hole)
* Media opacity will not be an exclusion criterion provided that the investigator can assess the presence or absence of DME on OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects avoiding 15 letters (3 lines) of best-corrected distance visual acuity loss at 18 weeks after cataract surgery. Distribution of visual acuity changes at 18 weeks after cataract surgery | 1 to 18 weeks post-cataract surgery
Distribution of absolute levels of distance visual acuity at 18 weeks after cataract surgery | 1 to 18 weeks post-cataract surgery
Analysis of time to 15 letter improvement of best-corrected distance visual acuity through 18 weeks after cataract surgery using a 2-state stochastic model to account for events and recoveries from events | 1 to 18 weeks post-cataract surgery

SECONDARY OUTCOMES:
Analysis of improvement of fluorescein leakage seen on fluorescein angiography at 18 weeks after cataract surgery | pre-cataract surgery to 18 weeks post-cataract surgery
Analysis of decrease in retinal thickness by OCT at 18 weeks after cataract surgery | pre-cataract surgery to 18 weeks post-cataract surgery
Analysis of level of diabetic retinopathy using recognized photographic grading system at 18 weeks after cataract surgery | pre-cataract surgery to 18 weeks post-cataract surgery
Additional changes 12 weeks after discontinuation of pegaptanib (6 months after study entry) | pre-cataract surgery to 6 months post-cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Oliver D. Schein, MD, MPH, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States